CLINICAL TRIAL: NCT04844047
Title: Does Fall Arrest Strategy Training (FAST) Added to a Fall Prevention Program Improve Physical Capacity to Prevent Serious Fall-related Injury in Older Women?
Brief Title: Does Fall Arrest Strategy Training Improve Capacity to Prevent Fall-Related Injury in Older Women?
Acronym: FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Cathy Arnold, Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BIO-REB 16-72
Record Dates: First submitted 2021-03-08; First posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Fall Injury
Keywords: fall risk; older adult; injury prevention
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors were blinded to intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAST (Active Comparator): Twice per week exercise program, 45 minutes duration for 12 weeks conducted in the community. Participants attended a 30-minute fall prevention education session once per week. FAST followed the same principles as Standard, with the addition of the following goals: 1) Increase UE strength (shoulder girdle/arm) utilizing both concentric and eccentric contractions, 2) Improve trunk and neck postural control during slow and fast body motions, 3) Optimize forward descent strategies via practice of quick response reaching, landing and controlled descent with hands on the wall or on the floor as able. Training progression for strength and body control included increasing the distance standing from the wall, progressing to one arm descents, increasing reps and speed and moving to greater gravity and body weight resistance such as hands and knees position on the floor as able. Quick movement practice targeted unexpected reaching activities, balloon and ball toss
  Interventions: Other: Exercise
- Standard (Placebo Comparator): Twice per week exercise program, 45 minutes duration for 12 weeks conducted in a community site (assisted living residence). Participants also attended a 3o minute fall prevention education session once per week. The Standard intervention consisted of a fall prevention exercise program designed for community-dwelling older adults. Exercises focussed on balance, leg strength, walking and mobility exercises designed to decrease fall risk.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — refer to arm descriptors
  Other Names: FAST
  Arms: FAST
Other: Exercise — refer to arm descriptors
  Other Names: Standard
  Arms: Standard

SUMMARY:
Falls are the leading cause of injury hospitalization for seniors across Saskatchewan and addressing the underlying causes is a provincial health priority. Older women are more vulnerable to the most common fall-related injuries (upper body) during forward falling while walking. Exercise programs designed to improve balance and strength can reduce fall risk but it is not known if specific exercises targeted to upper body strength and agility can improve chances for safe landing when a fall is inevitable. The investigators have developed such a program, Fall Arrest Strategy Training (FAST) and successfully piloted the feasibility of the exercises to be included in a standard fall prevention program. FAST is meant to increase arm strength, reaction time, trunk control, and teach better landing techniques. The potential efficacy of such an intervention to improve landing capacity has not been studied in older women. Thirty-two women age 60 years or older will be randomly assigned to either FAST or a Standard Exercise group. Half will do standard exercises targeting balance, mobility and lower extremity strength; the other half will do the same exercises with the addition of FAST. Both groups will exercise twice per week for 12 weeks. Participants will be tested before and after for arm strength, reaction time, balance, mobility and the ability to control body descent (absorb energy) using a technique we developed in our lab. While in a safety harness, participants will simulate a forward fall onto a platform that measures energy during impact. While completely preventing falls is not possible, this study will help the investigators learn if simple exercises like FAST combined with balance training can decrease fall risk AND reduce the risk of serious injury when a fall is unavoidable. It will help address the growing personal and societal cost of fall-related injury. This study will also inform future research targeted to include a large-scale trial evaluating the impact and implementation of FAST training in older adults across the spectrum of care and development of a computer simulation model to determine which factors are most important for reducing the risk of fall-related injury.

DETAILED DESCRIPTION:
Falls are the current leading cause of fracture and head injury in older adults in Saskatchewan and will continue to be a growing health concern given the aging population. Determining effective and feasible interventions to prevent the downward spiral of failing health, admission to long term care and even death following a serious fall-related injury is important to Saskatchewan seniors, the health care team, policy makers and the public at large.

Exercise is known to decrease fall risk in community-dwelling older adults and should theoretically also reduce risk for injury during a fall; however, there are no clinical trials evaluating exercises designed specifically to enhance safe landing when a fall is imminent. Ideally, the health care team would like to support older adults in preventing all falls but in reality, this is not possible. Developing an intervention targeting both fall AND injury prevention (in the event a fall is inevitable) should enhance the effectiveness of exercise for reducing fall-related injury. This study will investigate the efficacy of novel Fall-Arrest Strategy Training (FAST) to improve the physical capacity to arrest a fall and reduce injury risk in older community-dwelling women.

The risk of injury from falls depends on both the severity of impact and neuromuscular capacity such as bone and muscle strength of the affected body part. Sixty percent of all falls in older adults occur in a forward direction, more often in women than men. Forward falls are typically combined with hand contact as a protective response to prevent head, hip or torso injury. The effectiveness of these important protective strategies unfortunately decreases with aging. Evidence suggests forward fall arrest strategies can be modified to improve safe landing and reduce impact forces. The critically important question is whether older adults, in particular older women at high risk for fracture, can enhance their ability to efficiently utilize fall arrest strategies intended to diminish both the risk of head impact and the risk of wrist fracture.

Fall Arrest Strategy Training (FAST) is a new, innovative exercise intervention the investigators have developed uniquely focusing on enhancing upper extremity (UE) strength, response time, trunk control and specific strategies to safely lower the body. The severity of impact with a forward fall is determined primarily by pre-impact neuromuscular factors - muscle strength, movement time, and kinematic placement of the upper extremity (UE) which may also depend on available joint range of motion (ROM). FAST uses functional exercises specifically targeted to address these factors and are easily incorporated into general fall prevention programs. Staying on Your Feet is an established and effective fall prevention program offered to community-dwelling older adults in the Saskatoon Health Region. The feasibility of implementing FAST into Staying on Your Feet was verified in a previous pilot study. The important extension of this work is to determine if functional improvements result in improved fall-specific neuromuscular capacity and ability to absorb energy. The focus of this project is to further advance our understanding of the effect of FAST on functional fall risk outcomes and fall-arrest capacity in older women.

The goal of FAST is to increase fall-arrest capacity, defined as neuromuscular ability that could be utilized to prevent and minimize injury during a fall. While fall-related injury risk is difficult to measure directly, increases in fall-arrest capacity will likely lead to a reduction in that risk. Therefore, the effectiveness of injury risk reduction interventions such as FAST can be measured by their ability to increase fall-arrest capacity. One important factor recently emerging in the falls literature is energy absorption; older women absorb less energy in their UE during a controlled forward descent compared to younger women. The investigators have developed an experimental apparatus which can measure UE energy absorption in both controlled and unexpected forward body descents. Muscle strength, particularly surrounding the shoulder girdle and elbow, is another important forward fall-arrest capacity factor.

The purpose of this study is to advance knowledge of this innovative and simple training program, FAST, integrated into fall prevention programming, to determine if it has potential to improve the physical capacity to arrest a fall and reduce injury risk in older community-dwelling women. This proposed study will use novel lab-based energy absorption and strength measures, combined with functional measures of mobility and fall risk. Fall-arrest capacity changes after an intervention such as FAST have never been examined in older women.

Research Goals and Objectives: The principal research questions of this study are: 1) Does the addition of FAST training lead to improvements in UE energy absorption during controlled and unexpected forward descents as compared to a Standard fall prevention exercise program (Standard Exercise) focusing on walking, balance and lower extremity strength? 2) Does FAST produce greater gains in functional arm muscle strength, response time, mobility and balance control compared to Standard Exercise? The hypotheses are that FAST will result in greater improvements in energy absorption, UE strength, response time and mobility compared to Standard Exercise at the end of 12 weeks of training with similar gains in fall risk and balance control.

Trial Design and Methodology: The proposed study is a pilot randomized trial where women, age 60 years or older living in the community will be randomly assigned to either FAST or Standard Exercise. Education on fall prevention will be provided to both groups. The exercise groups will be offered in the community, coordinated with an existing fall prevention program (Staying on Your Feet; Saskatoon Health Region). Participants will be recruited via announcements and posters in the community. Interested participants are invited to attend an information session prior to the start of the program and a screening questionnaire will be administered in person or by telephone. Eligibility criteria is explained in detail elsewhere. Eligible participants will be randomly assigned to either group using a random allocation conducted by someone not directly involved in the study. Measures will be collected at the College of Kinesiology Biomechanics of Balance and Movement Lab, University of Saskatchewan at the start of the training (baseline), and immediately post intervention. An experienced physical therapist or exercise therapist will supervise FAST and Standard Exercise. Both exercise programs will occur twice per week, 45 minutes duration, for 12 weeks at a community site. FAST will include the same exercises to improve balance, walking and general mobility as Standard Exercise, but will also incorporate FAST training.

Outcome Measures: Outcome measures are designed to inform five primary fall-arrest capacity variables: 1) energy absorption in controlled descent, 2) energy absorption in unexpected descent, 3) eccentric muscle strength, 4) concentric muscle strength, 5) UE response time and secondary measures of fall risk, joint range of motion and balance and are described in detail elsewhere.

Analysis: Effect sizes for this study were estimated using variability data from our previous fall-arrest capacity work with young and older women and other published UE energy data. Our pilot data with older adults has shown a 20% higher energy absorption in adults who perform more UE training. A clinically meaningful increase in energy absorption is unknown. Based on our data, a 25% increase in the energy absorption will require 16 participants per group to detect differences at 80% power. Intention-to-treat analysis will be conducted using all participants assigned to intervention or control sites. A completer only analysis (based on attendance rates) will also be conducted. Repeated measures MANOVA tests will test for time and time*group differences across the 12 week time period for the five primary variables: energy absorption in controlled an unexpected descent, concentric and eccentric arm muscle strength and UE reaction time as well as the secondary measures of joint mobility, balance and fall risk. Given the exploratory nature of this study, significance will be set at p<0.05 for omnibus tests.

ELIGIBILITY:
Inclusion Criteria:

- Women aged 60 years or older living in the community.

Exclusion Criteria:

* Any recent upper body (hand, wrist, shoulder, trunk, neck) injury or painful joint problem that limited day to day activities or resulted in pain on a daily basis,
* A prior distal radius fracture in the past 2 years,
* Any fracture in the past year, or multiple fractures of the wrist or forearm,
* Any history of UE neurological problems (i.e. Stroke, Multiple Sclerosis, Parkinson's Disease, Reflex Neuropathy),
* Any cardio-vascular problems that would contradict UE strength testing or training,
* Any signs of severe cognitive impairment or
* Unable to safely ambulate independently (with or without a walking aid) in the community.

A medical and demographic screening questionnaire as well as the Mini-Cog (Borson et al, 2000) were used to determine eligibility.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self identification as female is inclusion criteria
Enrollment: 40 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-04-18 (Actual)

PRIMARY OUTCOMES:
UE Strength - Isometric | 12 weeks
  Measured with a hand-held dynamometer; mean of three trials for shoulder abduction, shoulder flexion and elbow extension
UE Strength - Grip | 12 weeks
  Measured with a dynamometer; participant in sitting, standardized elbow flexion position and handle position, gripping maximum exertion; mean of three trials for shoulder abduction, shoulder flexion and elbow extension
UE Strength - Isometric Push-off Test | 12 weeks
  Measured with a hand-held dynamometer for grip strength with the handle inverted and stabilized on a table top. Participant pushes downward in a standing position; mean of 3 trials used
UE Strength - Isokinetic Concentric and Eccentric | 12 weeks
  Using a protocol developed in the investigators' lab, with the Humac Norm isokinetic dynamometer. An upper extremity pushing motion of primarily elbow extension measuring maximal force for concentric and eccentric motion. Mean of three trials used
UE Mobility | 12 weeks
  Shoulder Extension and Wrist Extension Active Range of Motion with passive overpressure measure with a manual goniometer in a sitting position
UE Response Time | 12 weeks
  Time from the start of an auditory cue to lift hands from a position standing with arms at side of body to the first touch on a force from auditory cue to touching a forceplate at shoulder level. Mean of three trials for right, left and both hands together used.
Balance - One Leg Standing | 12 weeks
  Timed ability to stand on one leg with no support, up to 60 seconds. Two trials on each leg
Balance - Tandem Standing | 12 weeks
  This is a standard test first described by Hile et al (2012) where the participant tries standing in a tandem position, one foot in front of the other first with and then without support for up to 30 seconds without support. Scored on a scale of 5, with maximum score of 5 meaning standing without support for full 30 seconds
Self Report Fall Risk - FROP-Com | 12 weeks
  Fall Risk for Older People living in the Community (National Aging Research Institute, 2012 http://www.mednwh.unimelb.edu.au/nari_tools/nari_tools_falls.html) measures fall risk in 13 categories, for a total possible score of 60 (higher risk)
Self Report Balance Confidence | 12 weeks
  Activities Balance Confidence Scale (ABC; Powell & Myers 1995) rating of confidence for 16 day to day functional tasks on a scale 0 - 100; mean of 16 items used as total score
Sit to Stand Test | 12 weeks
  Number of full sit to stand movements completed within 30 seconds with arms crossed. One practice followed by actual test
Timed Up and Go Test (TUG) | 12 weeks
  Timed test to stand up from a chair, walk 3 meters, turn to chair and sit down. One practice trial, followed by one timed test (Podsiadlo & Richardson 1991)
Ground Reaction Force | 12 weeks
  Forward Descent and Landing Apparatus used to measure a controlled and unexpected release onto outstretched hands (simulated forward fall). Bilateral force platforms recorded ground reaction forces as participants performed a controlled descent with body at an angle 30 degrees from vertical, and then in an unexpected release while tethered to the ceiling, shoulders in 90 degrees of flexion and hands just hovering above force plate. Mean of 3 trials.
Elbow ROM during simulated forward descent | 12 weeks
  Forward Descent and Landing Apparatus used to measure a controlled and unexpected release onto outstretched hands (simulated forward fall). An eight camera motion capture system collected 3D upper extremity kinematics. Maximal elbow ROM was measured as participants performed a controlled descent with body at an angle 30 degrees from vertical, and then in an unexpected release while tethered to the ceiling, shoulders in 90 degrees of flexion and hands just hovering above force plate. Mean of 3 trials.
Peak elbow moment and elbow stiffness during simulated forward descent | 12 weeks
  Forward Descent and Landing Apparatus used to measure a controlled and unexpected release onto outstretched hands (simulated forward fall). An eight camera motion capture system collected 3D upper extremity kinematics. Elbow moments and stiffness values were calculated, normalized to height and body weight. Participants performed a controlled descent with body at an angle 30 degrees from vertical, and then in an unexpected release while tethered to the ceiling, shoulders in 90 degrees of flexion and hands just hovering above force plate. Mean of 3 trials.
Energy Absorption during simulated forward descent | 12 weeks
  Forward Descent and Landing Apparatus used to measure a controlled and unexpected release onto outstretched hands (simulated forward fall). An eight camera motion capture system collected 3D upper extremity kinematics. Energy absorption was calculated calculated using the total ground reaction force and the movement of the shoulders as a measure of the vertical displacement of the body, normalized to height and body weight. Participants performed a controlled descent with body at an angle 30 degrees from vertical, and then in an unexpected release while tethered to the ceiling, shoulders in 90 degrees of flexion and hands just hovering above force plate. Mean of 3 trials.

SECONDARY OUTCOMES:
Falls | 64 weeks
  number of reported falls
Muscle Activity | 12 weeks
  EMG analysis of muscle activity during controlled and quick descents

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Arnold, PhD, Principal Investigator — School Of Rehabilitation Science, University Of Saskatchewan

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be disseminated. Participants will receive aggregate summary of findings and confidential individual information as requested

REFERENCES:
- [Background] DeGoede KM, Ashton-Miller JA. Fall arrest strategy affects peak hand impact force in a forward fall. J Biomech. 2002 Jun;35(6):843-8. doi: 10.1016/s0021-9290(02)00011-8. PMID 12021005
- [Background] DeGoede KM, Ashton-Miller JA. Biomechanical simulations of forward fall arrests: effects of upper extremity arrest strategy, gender and aging-related declines in muscle strength. J Biomech. 2003 Mar;36(3):413-20. doi: 10.1016/s0021-9290(02)00396-2. PMID 12594989
- [Background] Borson S, Scanlan J, Brush M, Vitaliano P, Dokmak A. The mini-cog: a cognitive 'vital signs' measure for dementia screening in multi-lingual elderly. Int J Geriatr Psychiatry. 2000 Nov;15(11):1021-7. doi: 10.1002/1099-1166(200011)15:113.0.co;2-6. PMID 11113982
- [Background] Sran MM, Stotz PJ, Normandin SC, Robinovitch SN. Age differences in energy absorption in the upper extremity during a descent movement: implications for arresting a fall. J Gerontol A Biol Sci Med Sci. 2010 Mar;65(3):312-7. doi: 10.1093/gerona/glp153. Epub 2009 Oct 27. PMID 19861641
- [Background] Lee Y, Ashton-Miller JA. The effects of gender, level of co-contraction, and initial angle on elbow extensor muscle stiffness and damping under a step increase in elbow flexion moment. Ann Biomed Eng. 2011 Oct;39(10):2542-9. doi: 10.1007/s10439-011-0308-3. Epub 2011 Apr 12. PMID 21484509
- [Background] Lo J, McCabe GN, DeGoede KM, Okuizumi H, Ashton-Miller JA. On reducing hand impact force in forward falls: results of a brief intervention in young males. Clin Biomech (Bristol). 2003 Oct;18(8):730-6. doi: 10.1016/s0268-0033(03)00124-4. PMID 12957559
- [Background] Maki BE, McIlroy WE. Control of rapid limb movements for balance recovery: age-related changes and implications for fall prevention. Age Ageing. 2006 Sep;35 Suppl 2:ii12-ii18. doi: 10.1093/ageing/afl078. PMID 16926197
- [Background] Public Health Agency of Canada. Seniors' Falls in Canada. 2nd Report. 2014; www.phac-aspc.gc.ca/seniors-aines [On-line].
- [Background] Schonnop R, Yang Y, Feldman F, Robinson E, Loughin M, Robinovitch SN. Prevalence of and factors associated with head impact during falls in older adults in long-term care. CMAJ. 2013 Nov 19;185(17):E803-10. doi: 10.1503/cmaj.130498. Epub 2013 Oct 7. PMID 24101612
- [Background] Sherrington C, Whitney JC, Lord SR, Herbert RD, Cumming RG, Close JC. Effective exercise for the prevention of falls: a systematic review and meta-analysis. J Am Geriatr Soc. 2008 Dec;56(12):2234-43. doi: 10.1111/j.1532-5415.2008.02014.x. PMID 19093923
- [Background] Chiu J, Robinovitch SN. Prediction of upper extremity impact forces during falls on the outstretched hand. J Biomech. 1998 Dec;31(12):1169-76. doi: 10.1016/s0021-9290(98)00137-7. PMID 9882050
- [Background] Arnold CM, Walker-Johnston J, Lanovaz JL, Lattimer LJ. Does Fall Arrest Strategy Training Added to a Fall Prevention Programme Improve Balance, Strength, and Agility in Older Women? A Pilot Study. Physiother Can. 2017;69(4):323-332. doi: 10.3138/ptc.2016-27EP. PMID 30369700
- [Background] Lattimer LJ, Lanovaz JL, Farthing JP, Madill S, Kim S, Robinovitch S, Arnold C. Female Age-Related Differences in Biomechanics and Muscle Activity During Descents on the Outstretched Arms. J Aging Phys Act. 2017 Jul;25(3):474-481. doi: 10.1123/japa.2016-0102. Epub 2017 Jun 28. PMID 28095094
- [Background] Lattimer LJ, Lanovaz JL, Farthing JP, Madill S, Kim SY, Robinovitch S, Arnold CM. Biomechanical and physiological age differences in a simulated forward fall on outstretched hands in women. Clin Biomech (Bristol). 2018 Feb;52:102-108. doi: 10.1016/j.clinbiomech.2018.01.018. Epub 2018 Feb 3. PMID 29407858